CLINICAL TRIAL: NCT04360278
Title: Plasma Collection From Convalescent and/or Immunized Donors for the Treatment of COVID-19
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200092; 20-CC-0092
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: Titer; Antibodies; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Plasma Donors: Persons who have recovered from COVID-19 or have been immunized against SARS-CoV-2 who meet criteria to donate plasma.

SUMMARY:
Background:

The Coronavirus disease 2019 (COVID-19) pandemic is a major public health issue. Researchers want to collect plasma from people who have recovered from COVID-19, and use this plasma to treat people who are sick with the disease. The plasma will have antibodies against the virus that causes COVID-19. Persons who have received a COVID-19 vaccine may also donate plasma that contains antibodies against the virus if they meet criteria according to the FDA.

Objective:

To collect plasma from people who have recovered from COVID-19 or have been vaccinated against the coronavirus that causes COVID-19, so that the plasma can be used to treat people with the disease.

Eligibility:

Adults ages 18 and older who have been diagnosed with, and have recovered from, COVID-19.

Design:

Participants will be screened with a physical exam, medical history, and blood sample. Their pulse, blood pressure, and temperature will be taken. Their height and weight will be recorded.

Participants will donate plasma. It will be collected through whole blood donation or through apheresis.

For whole blood donation, a needle will be placed in the participant s arm vein. Blood will be withdrawn.

For apheresis, a needle will be placed in the participant s arm vein. Blood will be withdrawn. A machine will separate the plasma from the red cells. The plasma will be removed, and the rest of the cells will be returned to the participant either through the same needle or through a needle in their other arm.

Participants will have 3 to 20 plasma donations.

Participation will last up to 3 years.

DETAILED DESCRIPTION:
Emerging infectious diseases such as the Coronavirus disease 2019 (COVID-19) pandemic cause substantial morbidity and mortality. During the early emergent phases of such diseases, there is often no vaccine to prevent infection, nor specific therapeutic agent to treat the disease. The objective of this protocol is the collection of immune plasma from persons post-recovery from COVID-19 or vaccination against SARS-CoV-2. This plasma may potentially be used in the treatment or prophylaxis of active COVID-19 under other protocols.

Candidates will be screened for eligibility to participate in plasma donations and their blood levels of antibodies to SARS-CoV-2. Enrolled subjects will receive a baseline physical and laboratory examination. Subjects with sufficient anti-SARS-CoV-2 antibody titers who meet standard blood bank criteria for plasma donation will then be scheduled for plasma collections. Plasmapheresis is the preferred method of collection, with up to 800 mL of plasma collected per donation depending on the weight of the donor. Collected immune plasma will be tested for blood-borne pathogens, and stored according to standard blood bank procedures. The scope of this protocol is limited to collection of plasma from subjects with sufficiently high anti-SARS-CoV-2 antibody titer. Any administration of convalescent immune plasma to subjects will be performed under a separate protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ability of subject to understand, ask questions, and the willingness to sign the written informed consent document
* Age >=18 years
* Ability to meet blood donor eligibility criteria as defined in the FDA Code of Federal Regulations 21 CFR 630, AABB Standards and DTM SOP, including:

  * Weight >=110 pounds (50 kg)
  * Adequate peripheral venous access for plasma donation (as judged by the examiner)
  * Vital signs (with exceptions as acceptable per DTM SOP)
* For COVID-19 convalescent subjects, the following criteria must be met:

  * Prior diagnosis of COVID-19 documented by a laboratory test or by physician attestation
  * Complete resolution of symptoms for at least 10 days prior to donation.
  * Donors with residual loss of taste/smell are acceptable as long as they have no acute symptoms of COVID-19
* For vaccinated subjects, the following criteria must be met:

  --Subjects must meet FDA donor eligibility criteria to donate convalescent plasma
* Willingness to engage in repeat plasma collections for a 120-day period with possible extension per FDA guidance, provided anti-SARS-CoV-2 titers remain sufficiently high
* Willingness to have samples stored for clinical and/or genetic research testing

EXCLUSION CRITERIA:

* Patients who cannot give proper informed consent due to inability to understand the nature of the proposed therapy and attendant risk
* Age under 18 years
* Females must not be pregnant (per routine blood donor criteria)
* Any sign of active infection, including but not limited to:

  * Subjective or documented fever (>37.5 (Infinite)C)
  * Cough
  * Shortness of breath
  * Diarrhea
* Antibiotics within the prior 48 hours
* Considered immune suppressed for example current use of oral or parenteral steroids, highdose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs
* Permanent deferral from blood donation as defined in the FDA Code of Federal Regulations 21 CFR 630, AABB Standards, and DTM SOP
* Participation in medical research outside DTM that includes:

  --Protocols that are currently ongoing or will start during the duration of this study that require more than 500 mL of blood to be given in any 8-week period of time
* Total plasma protein level < 6.0 g/dL
* Unwillingness to engage in repeat plasma collections for a 120-day period with possible extension per FDA guidance, provided anti-SARS-CoV-2 titers remain sufficiently high
* Unwillingness to have samples stored for clinical and/or genetic research testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community donors who have recovered from COVID-19, or have been immunized against SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Collection of convalescent plasma | 240 days
  Successful collection of convalescent or immunized donor plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Kamille A West-Mitchell, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.aa

REFERENCES:
- [Derived] Gedda MR, Danaher P, Shao L, Ongkeko M, Chen L, Dinh A, Thioye Sall M, Reddy OL, Bailey C, Wahba A, Dzekunova I, Somerville R, De Giorgi V, Jin P, West K, Panch SR, Stroncek DF. Longitudinal transcriptional analysis of peripheral blood leukocytes in COVID-19 convalescent donors. J Transl Med. 2022 Dec 12;20(1):587. doi: 10.1186/s12967-022-03751-7. PMID 36510222
- [Derived] De Giorgi V, West KA, Henning AN, Chen LN, Holbrook MR, Gross R, Liang J, Postnikova E, Trenbeath J, Pogue S, Scinto T, Alter HJ, Cantilena CC. Naturally Acquired SARS-CoV-2 Immunity Persists for Up to 11 Months Following Infection. J Infect Dis. 2021 Oct 28;224(8):1294-1304. doi: 10.1093/infdis/jiab295. PMID 34089610
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-CC-0092.html